CLINICAL TRIAL: NCT04308642
Title: Pilot Study to Evaluate Blood and Urine Kidney Injury Markers to Facilitate Early Detection of Renal Adverse Drug Events in Pediatric Cancer Patients Treated With Nephrotoxic Chemotherapy (Kid-MaCare Oncology)
Brief Title: Study to Evaluate Blood and Urine Kidney Injury Markers to Facilitate Early Detection of Renal Adverse Drug Events in Pediatric Cancer Patients Treated With Nephrotoxic Chemotherapy
Acronym: Kid-MaCareOnco
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Stiftung für Krebskranke Kinder (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-02143; ks19Pfister
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Kidney Impairment
Keywords: nephrotoxic chemotherapy; pediatric cancer patients; renal adverse drug events; renal function; renal tubular injury; Uromodulin; drug related kidney injury; kidney markers
MeSH Terms: conditions — Renal Insufficiency | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood test for renal biomarkers — blood test for renal biomarkers (uromodulin,Neutrophil gelatinase-associated lipocalin, beta-trace protein, creatinine, cystatin C)
Other: urine test for renal biomarkers — urine test for renal biomarkers (uromodulin, alpha-1 microglobulin, retinol-binding protein, Neutrophil gelatinase-associated lipocalin (NGAL), beta-trace protein, cylinder, albumin, immunoglobulin G (IgG), transferrin, creatinine)

SUMMARY:
This study is to investigate blood and urine kidney injury markers (especially Uromodulin) in pediatric cancer patients treated with nephrotoxic chemotherapy. Uromodulin is a marker to detect and monitor tubular injury and renal function.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent by their-selves (≥ 14 years) or their legal representatives (< 14 years or in case of lacking capacity of judgement)
* cancer diagnosis, that indicates a nephrotoxic chemotherapy including the drugs High Dose MTX (HD-MTX), ifosfamide, cis- and carboplatin.

Exclusion Criteria:

* critically-ill patients with inotropic and/or vasopressor drugs
* signs of severe Sepsis
* receiving other nephrotoxic drugs parallel to the chemotherapy cycle

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients aged 0-18 years treated at the hematology-oncology at the University Children's Hospital Basel (UKBB) with a cancer diagnosis, that indicates a nephrotoxic chemotherapy including the drugs High Dose MTX (HD-MTX), ifosfamide, cis- and carboplatin.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in serum uromodulin levels (ng/ml) | from baseline (i.e. prior to first nephrotoxic chemotherapy cycle) to post-baseline (i.e. at the end of the first nephrotoxic chemotherapy cycle exposure); depending on chemotherapy protocol (maximally 24 - 72 hours)
  Change in serum uromodulin levels (ng/ml)

SECONDARY OUTCOMES:
Change in serum uromodulin levels (ng/ml) | at baseline (i.e. prior to first nephrotoxic chemotherapy cycle) and post-baseline (i.e. before, dur-ing and at the end of each nephrotoxic chemotherapy cycle),maximally 6- 9 months
  Change in serum uromodulin levels (ng/ml)
Change in urine uromodulin levels (ng/ml) | at baseline (i.e. prior to first nephrotoxic chemotherapy cycle) and post-baseline (i.e. before, dur-ing and at the end of each nephrotoxic chemotherapy cycle), maximally 6- 9 months
  Change in urine uromodulin levels (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pfister, Prof MD, Principal Investigator — University Children's Hospital Basel (UKBB), University of Basel
Locations (1):
- University Children's Hospital Basel (UKBB), University of Basel, Basel, Switzerland